CLINICAL TRIAL: NCT00585013
Title: A Trial of Inhaled Nitric Oxide (NO) as an Anti-Inflammatory and Anti-Reperfusion Agent in the Treatment of Infants and Children Undergoing Cardiopulmonary Bypass for Repair of Congenital Heart Disease
Brief Title: Inhaled NO as an Anti-inflammatory and Anti-reperfusion Agent in Infants and Children Undergoing Cardiopulmonary Bypass
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Mallinckrodt (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CHECP1
Record Dates: First submitted 2007-12-20; First posted 2008-01-02 (Estimated); Results first posted 2015-11-04 (Estimated); Last update posted 2015-11-04 (Estimated); Status verified 2015-11

CONDITIONS: Congenital Heart Disease
Keywords: Inhaled Nitric Oxide (NO); Anti-inflammatory; Anti-reperfusion agent
MeSH Terms: conditions — Heart Defects, Congenital | interventions — Nitric Oxide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nitric Oxide Delivery Group (Experimental): Patients will receive standard care with the addition of NO gas. During cardiopulmonary bypass, NO at 20 ppm will be added to the sweep gas of the extracorporeal circuit. Following termination of cardiopulmonary bypass, inhaled NO will be discontinued.
  Interventions: Drug: Nitric Oxide
- Placebo (No Intervention): Placebo delivery of oxygen at standard dose.

INTERVENTIONS:
Drug: Nitric Oxide — Patients will receive standard care with the addition of NO gas. During cardiopulmonary bypass, NO at 20 ppm will be added to the sweep gas of the extracorporeal circuit. Following termination of cardiopulmonary bypass, inhaled NO will be discontinued.
  Other Names: NO gas
  Arms: Nitric Oxide Delivery Group

SUMMARY:
Each year, there are over 400,000 cardiac surgical operations performed in the United States; of which 10,000 are performed on children. These operations are made possible by the use of the heart-lung bypass machine, also known as cardiopulmonary bypass. This machine allows for the body to be supported while the heart is repaired. While this machine has been life saving, it has risks and can lead to a variety of complications.

One such complication results from the fact that the patient's blood is exposed to the foreign material of the machine, such as plastic tubing. In nearly all cases of cardiac surgery, this leads to a whole body response in the patient following the operation. This response, inflammation, is characterized by alterations in the function of the heart and lungs, fever, fluid retention, and bleeding disorders in the postoperative period. While this is usually temporary and self limiting, significant morbidity occurs in approximately 1-2% of cases where this inflammatory response is present. Additionally, children appear to be more susceptible to this response. This can lead to significant postoperative complications that are not associated with the actually surgical procedure performed on the heart.

The exact cause of this response is not fully understood. However, it is important to understand the triggers, timing, and pattern of this complex inflammatory response in order to modify or arrest it. Unlike other situations associated with this type of whole-body inflammatory reaction such as trauma or overwhelming infection, cardiac surgical teams have the advantage of knowing when the trigger will occur (i.e. during the cardiac operation) and hence have the opportunity for preemptive intervention in an effort to minimize the response. One such effort is the focus of this proposal.

Nitric oxide (NO) is a gas that has been used for years in the treatment of lung disease in infants. It has been life saving and safe. Recently, it has been investigated for its anti-inflammatory effects outside the lungs. We propose delivering NO to the source of the greatest inflammation in cardiac surgery, the cardiopulmonary bypass machine. It is our intention to show that in doing so; we can minimize the inflammation found in the first 24 hours following cardiac surgery in children. If we are correct, the reduction of this inflammation will result in less damage to other organs of the child's body and improved outcome following surgery.

DETAILED DESCRIPTION:
I. Hypothesis

Treatment of children during surgery employing cardiopulmonary bypass with inhaled, exogenous nitric oxide (iNO) delivered to the cardiopulmonary bypass circuit will:

1. Modulate ischemia/reperfusion injury
2. Influence endothelial dysfunction
3. Ameliorate the bypass-triggered systemic inflammatory response

II. Specific Aims

Three specific aims will test this hypothesis:

Delivery of iNO to the cardiopulmonary bypass circuit will result in a decrease in:

1. Measures of end-organ dysfunction often associated with CPB; pulmonary function, cardiac injury markers, serum creatinine, and neurologic injury markers.
2. Measures of inflammatory response, specifically IL-6 and TNFa via its antioxidant properties.
3. Platelet activation and aggregation leading to reduced transfusion requirements.

III. Introduction and Background

* Cardiopulmonary bypass leads to ischemia/reperfusion injury. One of the mediators of this injury is oxygen radical production. NO is known to bind oxygen radical species.
* Cardiopulmonary bypass leads to endothelial dysfunction. This is mediated through cell-free hemoglobin binding endogenous NO, as seen in sickle cell disease.
* Both of these factors, separately and in combination, perpetuate the inflammatory response triggered by CPB. NO affects this response by interfering with this process. Additionally, NO is known to affect neutrophil chemotaxis as well as platelet activation and aggregation, both of which further amplify the inflammatory response.

IV. Basic Protocol Experimental Design In a prospective, randomized, controlled, blinded pilot trial we will compare 20 ppm of iNO delivered to the CPB circuit. Our study will target children undergoing cardiopulmonary bypass (CPB) for surgery for the correction of transposition of great arteries (TGA) and Tetralogy of Fallot (TOF).

Subjects Inclusion Undergoing repair of TGA and TOF < 16 years of age Exclusion Age > 16 years of age Pregnancy Known bleeding disorder

Treatment Protocol Following informed consent, blood will be drawn pre-operatively for baseline characteristics (methemoglobin, venous saturation, CBC, S100, gene expression profiles, BNP, cTnI, IL-6, IL-8, lactate, TNFalpha)[Table, Blood sample for Study]. Intra-operatively we will use a standardized anesthetic protocol unless contraindicated by specific patient clinical characteristics. Intraoperative measurements will include: aortic cross clamp time, and total cardiopulmonary bypass time. Intraoperative hemodynamic measurements will include: mean systemic blood pressure (MAP), central venous pressure, right atrial pressure pulmonary artery pressure, and pulmonary capillary wedge pressure (when available). Blood samples will be drawn following CPB upon arrival to the ICU and will be analyzed as above. Repeat blood samples for each will be drawn again after 12, 24, and 48 hours. Patients will be followed to the time of discharge. Ventilator settings, length of ICU and hospital stay will be recorded. All measurements in both groups will be the same. Time points will be referenced from the time of admission to the PICU for both groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients with the following congenital heart lesions who require cardiopulmonary bypass for surgical repair or palliation will be eligible:
* D-transposition of the great vessels (D-TGA)
* Tetralogy of Fallot (TOF)
* Children of age less than 16 years

Exclusion Criteria:

* Signs of persistently elevated pulmonary vascular resistance preoperatively
* Cardiac arrest one week prior to surgery
* Prior surgical procedure that required use of cardio-pulmonary bypass
* Acute or chronic infection such as sepsis or wound infections
* History of any pulmonary condition such as pneumonia or respiratory distress syndrome
* Patients that have received steroid treatment within the last month
* DiGeorge syndrome
* Active bleeding disorder
* Any other condition associated with non-cardiac morbidity
* Use of another investigational drug
* Age over 16 years.

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 17 (Actual)
Dates: Start 2008-01; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Checchia, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- St. Louis Children's Hospital, St Louis, Missouri, United States

REFERENCES:
- [Derived] Checchia PA, Bronicki RA, Muenzer JT, Dixon D, Raithel S, Gandhi SK, Huddleston CB. Nitric oxide delivery during cardiopulmonary bypass reduces postoperative morbidity in children--a randomized trial. J Thorac Cardiovasc Surg. 2013 Sep;146(3):530-6. doi: 10.1016/j.jtcvs.2012.09.100. Epub 2012 Dec 8. PMID 23228403

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were randomized by the research perfusionist using sequentially ordered randomization codes. The randomization codes were generated using a computerized random number generator. The entire care team was blinded to the delivery device and drug delivery. Only the study perfusionist was aware of randomization and delivery.
Pre-assignment Details: Seventeen patients consented and were enrolled in the study. There were eight consent failures. One patient was disqualified after consent and randomization due to intraoperative findings of a lesion inconsistent with preoperative diagnosis and change in operative plan.
Groups:
- 1 Treatment: Patients will receive standard care with the addition of NO gas. During cardiopulmonary bypass, NO at 20 ppm will be added to the sweep gas of the extracorporeal circuit. Following termination of cardiopulmonary bypass, inhaled NO will be discontinued.
  Nitric Oxide : Patients will receive standard care with the addition of NO gas. During cardiopulmonary bypass, NO at 20 ppm will be added to the sweep gas of the extracorporeal circuit. Following termination of cardiopulmonary bypass, inhaled NO will be discontinued.
- 2 Placebo: Placebo delivery of oxygen at standard dose.
Period: Overall Study
Arm/Group | 1 Treatment | 2 Placebo
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1 Treatment | 2 Placebo | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 8 | 8 | 16
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | .4 (.1) | .4 (.1) | .4 (.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 5
  Male | 7 | 4 | 11
Region of Enrollment [Number; unit: participants]
  United States | 8 | 8 | 16

OUTCOME MEASURES:

1. Primary Outcome: Serum Inflammatory Mediators Post CPB
Description: Inflammation measured through the measurement inflammatory mediators, serum interleukin-6, serum interleukin-8, and tumor necrosis factor. Baseline (preoperative, 0h, 12h, 24h, and 48h.
Time Frame: 48 hours
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Nitric Oxide Delivery Group | Placebo
Number analyzed (Participants) | 8 | 8
ng/mL
  Interleukin-6 Preoperative | 3.8 (3.5) | 3.4 (2.5)
  Interleukin-6, 0 hrs | 90.9 (44.6) | 78.3 (45.7)
  Interleukin-6, 12 hrs | 51.5 (38.7) | 73.3 (67.0)
  Interleukin-6, 24 hrs | 64.2 (28.4) | 80.7 (82.1)
  Interleukin-6, 48 hrs | 31.2 (30.6) | 39.4 (48.9)
  Interleukin-8, Preoperative | 60.9 (28.8) | 39.8 (39.0)
  Interleukin-8, 0 hrs | 189.8 (104.1) | 248.9 (191.7)
  Interleukin-8, 12 hrs | 144 (133.4) | 85.9 (59.9)
  Interleukin-8, 24 hrs | 101.5 (62.7) | 139.2 (162.1)
  Interleukin-8, 48 hrs | 134.2 (107.0) | 60.4 (33.7)
  Tumor Necrosis Factor Preoperative | 2.9 (0.8) | 3.2 (1.1)
  Tumor Necrosis Factor, 0 hrs | 3.2 (1.5) | 4.1 (1.6)
  Tumor Necrosis Factor, 12 hrs | 1.7 (0.07) | 1.9 (1.1)
  Tumor Necrosis Factor, 24 hrs | 1.7 (1.3) | 3.2 (2.9)
  Tumor Necrosis Factor, 48 hrs | 2.8 (0.09) | 2.1 (1.2)
Statistical Analysis 1: Comparison: Nitric Oxide Delivery Group vs Placebo; Test type: Superiority or Other; p > 0.05, Wilcoxon (Mann-Whitney) — This p value applies to all time points for all variables

2. Primary Outcome: Myocardial Injury
Description: Troponin levels correlate with myocardial injury. Greater troponin levels represent greater myocardial injury
Time Frame: 48 hours
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | 1 Treatment | 2 Placebo
Number analyzed (Participants) | 8 | 8
ng/mL
  Preoperative | 0.07 (0.07) | 0.06 (0.1)
  0 h | 50.6 (37.8) | 54.1 (15.5)
  12 h | 11.7 (3.2) | 15.9 (3.5)
  24 h | 8.9 (2.6) | 12.5 (2.7)
  48 h | 4.8 (1.6) | 7.6 (2.0)
Statistical Analysis 1: Comparison: 1 Treatment vs 2 Placebo; Test type: Superiority or Other; p > 0.05, Wilcoxon (Mann-Whitney) — This applies for measurements at preoperative and 0 h time points
Statistical Analysis 2: Comparison: 1 Treatment vs 2 Placebo; Test type: Superiority or Other; p < 0.05, Wilcoxon (Mann-Whitney) — This applies to measurements at time points 12 h, 24 h, and 48 h

3. Primary Outcome: Myocardial Function as Measured by B-type Natiuretic Peptide (BNP) Levels
Description: BNP levels correlate to ventricular and myocardial performance, function, and strain. Higher values represent greater strain and decreased function.
Time Frame: 48 hours
Measure: Mean (Standard Deviation); unit: pg/dL
Arm/Group | 1 Treatment | 2 Placebo
Number analyzed (Participants) | 8 | 8
pg/dL
  Preoperative | 24 (22) | 100 (195)
  0 h | 43 (34) | 94 (100)
  12 h | 494 (222) | 812 (300)
  24 h | 425 (154) | 938 (511)
  48 h | 558 (535) | 1298 (827)
Statistical Analysis 1: Comparison: 1 Treatment vs 2 Placebo; Test type: Superiority or Other; p > 0.05, Wilcoxon (Mann-Whitney) — This applies to measurements at preoperative, 0 h, and 48 h time points
Statistical Analysis 2: Comparison: 1 Treatment vs 2 Placebo; Test type: Superiority or Other; p < 0.05, Wilcoxon (Mann-Whitney) — This applies to time points at 12 h and 24 h

4. Primary Outcome: Ischemic Injury as Measured by Lactate Levels
Description: Lactate levels correlate to ischemic injury. Higher values represent more injury.
Time Frame: 48 hours
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | 1 Treatment | 2 Placebo
Number analyzed (Participants) | 8 | 8
mmol/L
  Preoperative | 0.9 (0.2) | 0.5 (0.1)
  0 h | 1.9 (0.6) | 1.9 (1.0)
  12 h | 1.5 (0.4) | 1.5 (0.5)
  24 h | 1.4 (0.5) | 1.4 (0.4)
  48 h | 1.1 (0.2) | 1.1 (0.2)
Statistical Analysis 1: Comparison: 1 Treatment vs 2 Placebo; Test type: Superiority or Other; p > 0.05, Wilcoxon (Mann-Whitney) — Applies to all time points

5. Secondary Outcome: Incidence of Methhemoglobin >5%, Gene Expression Profiles, and S100B.
Time Frame: 48 hours
Population: Data not collected for these assessments
Arm/Group | 1 Treatment | 2 Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected throughout the hospital admission or to 30 days postoperative; whichever is longer.
Arm/Group | 1 Treatment | 2 Placebo
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/8 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No